CLINICAL TRIAL: NCT00245635
Title: Fluoxetine in Pediatric Body Dysmorphic Disorder
Acronym: FDA BDD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Eric Hollander, Prof. Psychiatry & Behavioral Sciences, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-10-302; 7R01FD002613-04 (FDA); NCT00029471 (obsolete NCT alias)
Record Dates: First submitted 2005-10-26; First posted 2005-10-28 (Estimated); Results first posted 2015-06-29 (Estimated); Last update posted 2018-04-27 (Actual); Status verified 2018-03

CONDITIONS: Body Dysmorphic Disorder
Keywords: Body Dysmorphic Disorder; BDD; BDD treatment; delusionality variant; OCD
MeSH Terms: conditions — Body Dysmorphic Disorders | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Fluoxetine (Experimental): Fixed/flexible dosing regimen of fluoxetine based on weight of subject and reaction to dosage, varying between 10mg and 80mg tablets once a day.
  Interventions: Drug: Fluoxetine
- Placebo (Placebo Comparator): Placebo tablets will be given 1/day for the duration of the study with a dosing schedule equivalent to that of the drug.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluoxetine — Tablets varying between 10mg and 80mg on a fixed/flexible dosing schedule based on the subjects' weight and side effects score.
  Other Names: Prozac
  Arms: Fluoxetine
Drug: Placebo — Placebo tablets will be given 1x/day for the duration of the study at a fixed/flexible dosing schedule similar to that for the drug fluoxetine based off of subjects' weight and side effects score.
  Arms: Placebo

SUMMARY:
This trial will study the effectiveness of the medication fluoxetine for children and adolescents ages 16 and younger with BDD who qualify.

DETAILED DESCRIPTION:
BDD usually begins in childhood or adolescence, but its treatment in pediatric populations has not been investigated. Recent data suggests that adults with BDD may respond to serotonin reuptake inhibitors (SRIs) such as fluoxetine (Prozac). Preliminary findings from case reports suggest that SRIs may also be effective in the treatment of BDD in children and adolescents. This study is the first large-scale, double-blind, placebo-controlled medication trial of fluoxetine for children and adolescents with BDD. Participants should be aged 16 or younger. Participation in this trial will last approximately 14 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female children and adolescents aged 16 and younger
* BDD or its delusional variant present currently and for at least 6 months prior to the study
* Ability to communicate meaningfully with the investigators and competent to provide written assent

Exclusion Criteria:

* Presence of Schizophrenia or Bipolar Disorder
* Recent suicide attempt or suicidal ideations that warrant hospitalizations
* Previous allergic reaction to fluoxetine
* History of a seizure disorder

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2004-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hollander, MD, Principal Investigator — Montefiore Medical Center/Albert Einstein College of Medicine
Locations (2):
- United States (2):
  - Montefiore Medical Center, Albert Einstein College of Medicine, The Bronx, New York
  - Rhode Island Hospital, Providence, Rhode Island

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fluoxetine | Placebo
Started | 25 | 18
Completed | 25 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluoxetine | Placebo | Total
Number analyzed (Participants) | 25 | 18 | 43
Age, Continuous [Mean (Full Range); unit: years] | 15.04 [9 to 18] | 14.88 [10 to 18] | 14.96 [9 to 18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 15 | 33
  Male | 7 | 3 | 10
Region of Enrollment [Number; unit: participants]
  United States | 25 | 18 | 43
BDD-Y-BOCS [Mean (Standard Deviation); unit: units on a scale] — Total scores at Baseline on the Body Dysmorphic Disorder-Yale-Brown Obsessive Compulsive Scale (BDD-Y-BOCS)
  units on a scale | 30.84 (4.2) | 35.16 (5.10) | 32.65 (5.02)

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Score on the BDD-Y-BOCS Scale
Description: To assess the change in total score on the Body Dysmorphic Disorder-Yale-Brown Obsessive Compulsive Scale (BDD-Y-BOCS) from baseline (visit 0) to endpoint (week 12). This is a 12-item scale that assesses obsessions and compulsions related to the patient's BDD. Each item's score ranges from 0 to 4, with a total possible score of 48 on the full assessment. Scores of 0 indicate no impairment, while scores of 4 indicate maximum impairment. Thus higher scores are considered to be a worse outcome.
Time Frame: Baseline compared to the study endpoint (week 12) [two time points]
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fluoxetine | Placebo
Number analyzed (Participants) | 25 | 18
units on a scale | -12.27 (11.78) | -9.53 (12.07)

ADVERSE EVENTS:
Time Frame: Adverse Event data was collected throughout the course of the study.
Description: Documentation of AE's were supplemented by checklists including the Fluoxetine Side Effects Scale and the SMURF.
Arm/Group | Fluoxetine | Placebo
Serious Adverse Events (participants affected / at risk) | 1/25 | 0/18
Other Adverse Events (participants affected / at risk) | 2/25 | 3/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluoxetine (N=25) | Placebo (N=18)
Suicidal Behavior (Psychiatric disorders) | 1 (1) | 0 (0) — Suicidal behavior was seen in one subject and had a possible relationship to study drug, and subject was seen in a partial hospitalization setting. This was reported to the IRB, FDA and DSMB.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluoxetine (N=25) | Placebo (N=18)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Weight Loss (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Trouble Sleeping (Nervous system disorders) | 1 (1) | 1 (1)
Nightmares (Nervous system disorders) | 1 (1) | 1 (1)
Stomach Pains (Gastrointestinal disorders) | 2 (2) | 1 (1)
Insomnia (Nervous system disorders) | 1 (2) | 0 (0)
Fatigue (General disorders) | 1 (3) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (2) | 2 (2)
Sweating (Endocrine disorders) | 1 (1) | 1 (1)
Agitated/Restlessness (Psychiatric disorders) | 1 (1) | 2 (2)
Dry Mouth (General disorders) | 1 (1) | 1 (1)
Silliness/Feeling too happy (Psychiatric disorders) | 1 (2) | 0 (0)
Headache (General disorders) | 1 (1) | 2 (2)
Lit Paper on Fire (Social circumstances) | 1 (1) | 0 (0)
Emotional (Psychiatric disorders) | 1 (1) | 0 (0)
Menstrual Cramps (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Forgetfulness (Psychiatric disorders) | 0 (0) | 1 (1)
Light hurts eyes (Eye disorders) | 0 (0) | 2 (2)
Feeling tense (Psychiatric disorders) | 0 (0) | 2 (2)
Ears ringing (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Drowsiness (General disorders) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Blurred/double Vision (Eye disorders) | 0 (0) | 2 (2)
Visit to ER: Family Conflict (Social circumstances) | 0 (0) | 1 (1)
Visit to ER: Aches (General disorders) | 0 (0) | 1 (1)
Itchiness (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Leg Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hair Loss (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Delay in Urination (Renal and urinary disorders) | 0 (0) | 1 (1)
Numbness (Nervous system disorders) | 0 (0) | 1 (1) — Hands and feet.
Tingling (Nervous system disorders) | 0 (0) | 1 (1) — Hands and Feet
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Heart Pounding/Racing (Cardiac disorders) | 0 (0) | 1 (2)
Trouble Keeping Balance (Nervous system disorders) | 0 (0) | 1 (1)
Room Spinning (Nervous system disorders) | 0 (0) | 1 (1)
Weight Gain (Metabolism and nutrition disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes